CLINICAL TRIAL: NCT01802333
Title: A Randomized Phase III Study of Standard Cytarabine Plus Daunorubicin (7+3) Therapy or Idarubicin With High Dose Cytarabine (IA) Versus IA With Vorinostat (NSC-701852) (IA + V) in Younger Patients With Previously Untreated Acute Myeloid Leukemia (AML)
Brief Title: Cytarabine and Daunorubicin Hydrochloride or Idarubicin and Cytarabine With or Without Vorinostat in Treating Younger Patients With Previously Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2013-00490; NCI-2013-00490 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1203; PS1203_A06PAMDREVW01; SWOG-S1203; S1203 (Other: SWOG); S1203 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; Idarubicin; Vorinostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (standard dose cytarabine, daunorubicin hydrochloride) (Experimental): INDUCTION/RE-INDUCTION: Patients receive standard dose cytarabine IV continuously on days 1-7 and daunorubicin hydrochloride IV on days 1-3. Patients with residual blasts may receive re-induction treatment beginning on day 15. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
  CONSOLIDATION: Patients receive cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5.
  TRANSPLANT: Patients may undergo an allogeneic transplant after induction therapy or consolidation therapy.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Other: Laboratory Biomarker Analysis
- Arm II (high-dose cytarabine, idarubicin) (Experimental): INDUCTION/RE-INDUCTION: Patients receive high dose cytarabine IV continuously on days 1-4 and idarubicin IV over 15 minutes on days 1-3. Patients with residual blasts may receive re-induction treatment beginning on day 28. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
  CONSOLIDATION: Patients receive cytarabine IV continuously on days 1-3 and idarubicin IV over 15 minutes on days 1-2.
  TRANSPLANT: Patients may undergo an allogeneic transplant after induction therapy or consolidation therapy.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cytarabine; Drug: Idarubicin; Other: Laboratory Biomarker Analysis
- Arm III (vorinostat, high-dose cytarabine, idarubicin) (Experimental): INDUCTION/RE-INDUCTIONI: Patients receive vorinostat PO TID on days 1-3, high-dose cytarabine IV continuously on days 4-7, and idarubicin IV over 15 minutes on days 4-6. Patients with residual blasts may receive re-induction treatment beginning on day 28. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
  CONSOLIDATION: Patients receive vorinostat PO TID on days 1-3, cytarabine IV continuously on days 4-6, and idarubicin IV over 15 minutes on days 4-5.
  TRANSPLANT: Patients may undergo an allogeneic transplant after induction therapy or consolidation therapy. (Permanently closed to accrual, effective 6/2/2015) Patients previously randomized to Arm III may continue treatment with or without vorinostat.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cytarabine; Drug: Idarubicin; Other: Laboratory Biomarker Analysis; Drug: Vorinostat

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic transplant
  Other Names: Allogeneic Hematopoietic Cell Transplantation; allogeneic stem cell transplantation; HSC; HSCT
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
  Arms: Arm I (standard dose cytarabine, daunorubicin hydrochloride)
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR
  Arms: Arm II (high-dose cytarabine, idarubicin); Arm III (vorinostat, high-dose cytarabine, idarubicin)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza
  Arms: Arm III (vorinostat, high-dose cytarabine, idarubicin)

SUMMARY:
This randomized phase III trial studies cytarabine and daunorubicin hydrochloride or idarubicin and cytarabine with or without vorinostat to see how well they work in treating younger patients with previously untreated acute myeloid leukemia. Drugs used in chemotherapy, such as cytarabine, daunorubicin hydrochloride, idarubicin, and vorinostat, work in different ways to stop the growth of cancer cells, either by killing the cells, stopping them from dividing, or by stopping from spreading. Giving more than one drug (combination chemotherapy) and giving the drugs in different doses and in different combinations may kill more cancer cells. It is not yet known which combination chemotherapy is more effective in treating acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare event-free survival (EFS) between patients with acute myeloid leukemia (AML) who receive standard 7+3 (cytarabine and daunorubicin hydrochloride) or idarubicin and high-dose cytarabine (IA) to patients who receive IA + vorinostat. (Chemotherapy) II. To determine whether it is possible to get 60% or more of adults with high-risk AML (by cytogenetics) in first complete remission (CR1) to allogeneic hematopoietic cell transplantation (HCT). (Transplant)

SECONDARY OBJECTIVES:

I. To estimate the frequency and severity of toxicities of the three regimens in this patient population. (Chemotherapy) II. To estimate disease-free survival (DFS) among patients who receive transplant. (Transplant) III. To compare event-free survival (EFS) between patients who receive standard 7 + 3 to patients who receive IA. (Chemotherapy) IV. To estimate the prevalence of the mutations nucleophosmin (nucleolar phosphoprotein B23, numatrin) (NPM1), isocitrate dehydrogenase 1 (NADP+), soluble (IDH1), isocitrate dehydrogenase 2 (NADP+), mitochondrial (IDH2), tet methylcytosine dioxygenase 2 (TET2) and deoxyribonucleic acid (DNA) (cytosine-5-)-methyltransferase 3 alpha (DNMT3A) and the cytogenetic risk distribution of patients on this study and to evaluate the association between these and overall survival (OS), event-free survival (EFS), disease-free survival (DFS), and complete remission rate. (Chemotherapy/Translational Medicine) V. To compare the complete response rate, disease-free survival (DFS), and overall survival (OS) between patients who receive standard 7+3 therapy or IA to patients who receive IA + vorinostat. (Chemotherapy)

TERTIARY OBJECTIVES:

I. Future planned studies will include testing of histone H3 acetylation, induction of gamma H2A histone family, member X (H2AX), analysis of reactive oxygen species (ROS) resistance and DNA methylation profiles. (Chemotherapy/Translational Medicine)

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

INDUCTION/RE-INDUCTION:

ARM I: Patients receive standard dose cytarabine intravenously (IV) continuously on days 1-7 and daunorubicin hydrochloride IV on days 1-3. Patients with residual blasts may receive re-induction treatment beginning on day 15. Patients achieving complete remission (CR) or complete remission with incomplete platelet recover (CRi) may proceed to allogeneic hematopoietic stem cell transplant (HSCT) or to consolidation therapy.

ARM II: Patients receive high dose cytarabine IV continuously on days 1-4 and idarubicin IV over 15 minutes on days 1-3. Patients with residual blasts may receive re-induction treatment beginning on day 28. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.

ARM III: Patients receive vorinostat orally (PO) thrice daily (TID) on days 1-3, high-dose cytarabine IV continuously on days 4-7, and idarubicin IV over 15 minutes on days 4-6. Patients with residual blasts may receive re-induction treatment beginning on day 28. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy. (Permanently closed to accrual, effective 6/2/2015) Patient previously randomized to Arm III may continue treatment without vorinostat.

CONSOLIDATION:

ARM I: Patients receive cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5.

ARM II: Patients receive cytarabine IV continuously on days 1-3 and idarubicin IV over 15 minutes on days 1-2.

ARM III: Patients receive vorinostat PO TID on days 1-3, cytarabine IV continuously on days 4-6, and idarubicin IV over 15 minutes on days 4-5. (Permanently closed to accrual, effective 6/2/2015) Patient previously randomized to Arm III may continue treatment with or without vorinostat.

In all arms, treatment repeats every 28 days for 4 courses or until transplant in the absence of disease progression or unacceptable toxicity.

TRANSPLANT: Patients may undergo an allogeneic transplant after induction therapy or consolidation therapy.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 - INDUCTION/RE-INDUCTION
* Patients must have morphologically confirmed newly diagnosed acute myelogenous leukemia (AML) with blood or bone marrow disease; patients with only extramedullary disease in the absence of bone marrow or blood involvement are not eligible; note: this protocol uses World Health Organization (WHO) diagnostic criteria for AML; patients with acute promyelocytic leukemia (APL, French-American-British [FAB], M3) or blastic transformation of chronic myelogenous leukemia (CML) are not eligible; patients with known core binding factor (CBF) or fms-like tyrosine kinase 3 (FLT3) related leukemias are eligible for this study, but should preferentially be placed on National Cancer Institute (NCI)-sponsored protocols specific for these subtypes, if available
* Patients must have diagnostic/pre-treatment specimens obtained within 28 days prior to registration submitted for cytogenetic (and fluorescent in situ hybridization [FISH] if possible) analysis to determine risk status; high risk classification will be defined as del(5q)/-5, del(7q)/-7, abn3q26 [inv(3)/t(3;3)], 11q23 rearrangement [except t(9;11)], 17p-, t(6;9), t(9;22), complex (at least 3 unrelated abnormalities [abn]), and monosomal karyotype (either loss of two different chromosomes or loss of one chromosome along with a structural chromosome abnormality other than add, ring and mar); karyograms and cytogenetics/FISH analysis reports must be submitted for discipline review
* Patients must be chemo-naïve, i.e., not have received any prior induction chemotherapy for AML or myelodysplastic syndrome (MDS); temporary prior measures such as apheresis or hydroxyurea are allowed; prior anthracycline therapy is allowed, but must not exceed a dose of 200 mg/m^2 daunorubicin or equivalent; prior all-trans retinoic acid (ATRA) for suspected APL is allowed; prior methotrexate for central nervous system (CNS) involvement is allowed; patients with prior history of MDS must not have received azacitidine, decitabine, lenalidomide or vorinostat
* Patients must have peripheral blood and bone marrow aspirate specimens obtained within 28 days prior to registration submitted for translational medicine; with patient consent, residuals will be banked for future research
* Patients must have Zubrod performance status =< 3
* Patients must have either echocardiogram (ECHO) or multi gated acquisition scan (MUGA) with ejection fraction >= 45% within 28 days prior to registration
* Patients must not have prolonged corrected QT (QTc) interval (> 500 msec) determined by electrocardiogram (EKG) within 28 days prior to registration
* Patients must not have cardiac disease defined as: New York Heart Association (NYHA) > class II; patients must not have unstable angina (angina symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Patients must not have any coexisting medical condition that is likely to interfere with study procedures or results, and must be reasonable candidates for intensive chemotherapy, in the opinion of their treating physicians
* Patients who are known to be human immunodeficiency virus (HIV) positive (+) are eligible providing they meet all of the following additional criteria within 28 days prior to registration:

  * Cluster of differentiation (CD) 4 cells >= 500/mm^3
  * Viral load < 50 copies of HIV messenger ribonucleic acid (mRNA)/mm^3 if on combination antiretroviral therapy (cART) or < 25,000 copies of HIV mRNA if not on cART
  * No zidovudine or stavudine as part of cART; patients who are HIV+ and do not meet all of these criteria are not eligible for this study
* Patients with known hepatitis B or hepatitis C infection may be eligible providing they have viral load < 800,000 IU/mL within 28 days prior to registration
* Patients must be able to take oral medications
* Patients must have a history and physical examination obtained within 28 days prior to registration
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Prior malignancy is allowed providing it does not require concurrent therapy; exception: active hormonal therapy is allowed
* Patients must not be receiving valproic acid
* All patients must be informed of the investigational nature of this study; patients or a legally authorized representative must sign and give written informed consent in accordance with institutional and federal guidelines
* As part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* STEP 2 - CONSOLIDATION
* Patients may be registered for consolidation provided that they were eligible for the initial induction/re-induction registration and satisfy the following additional criteria:

  * Patients must have achieved morphologic remission (complete remission [CR] or complete remission with incomplete blood count recover [CRi]) after completion of induction or re-induction therapy; patient must remain in remission until beginning consolidation and this must be documented by bone marrow and peripheral blood examination within 28 days prior to registration to Step 2
  * All non-hematologic treatment related toxicities that are deemed clinically significant by the treating physician must have resolved to =< grade 2
  * Patients must not have received allogeneic stem cell transplant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 754 (Actual)
Dates: Start 2013-02-12; Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — SWOG Cancer Research Network
Locations (447):
- United States (441):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Yuma Cancer Center, Yuma, Arizona
  - Mercy Cancer Center-Hot Springs, Hot Springs, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Assarian Cancer Center, Novi, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hemotology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Northwell Health/Center for Advanced Medicine, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Mountain Radiation Oncology, Asheville, North Carolina
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Transylvania Regional Hospital, Brevard, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Angel Medical Center, Franklin, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - McDowell Hospital, Marion, North Carolina
  - Blue Ridge Regional Hospital, Spruce Pine, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Derived] Garcia-Manero G, Podoltsev NA, Othus M, Pagel JM, Radich JP, Fang M, Rizzieri DA, Marcucci G, Strickland SA, Litzow MR, Savoie ML, Medeiros BC, Sekeres MA, Lin TL, Uy GL, Powell BL, Kolitz JE, Larson RA, Stone RM, Claxton D, Essell J, Luger SM, Mohan SR, Moseley A, Appelbaum FR, Erba HP. A randomized phase III study of standard versus high-dose cytarabine with or without vorinostat for AML. Leukemia. 2024 Jan;38(1):58-66. doi: 10.1038/s41375-023-02073-x. Epub 2023 Nov 7. PMID 37935977

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride): INDUCTION/RE-INDUCTION: Patients receive standard dose cytarabine IV continuously on days 1-7 and daunorubicin hydrochloride IV on days 1-3. Patients with residual blasts may receive re-induction treatment beginning on day 15. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
  CONSOLIDATION: Patients receive cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5.
  TRANSPLANT: Patients may undergo an allogeneic transplant after induction therapy or consolidation therapy.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic transplant
  Cytarabine: Given IV
  Daunorubicin Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Arm II (High-dose Cytarabine, Idarubicin): INDUCTION/RE-INDUCTION: Patients receive high dose cytarabine IV continuously on days 1-4 and idarubicin IV over 15 minutes on days 1-3. Patients with residual blasts may receive re-induction treatment beginning on day 28. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
  CONSOLIDATION: Patients receive cytarabine IV continuously on days 1-3 and idarubicin IV over 15 minutes on days 1-2.
  TRANSPLANT: Patients may undergo an allogeneic transplant after induction therapy or consolidation therapy.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic transplant
  Cytarabine: Given IV
  Idarubicin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Arm III (Vorinostat, High-dose Cytarabine, Idarubicin): INDUCTION/RE-INDUCTION: Patients receive vorinostat PO TID on days 1-3, high-dose cytarabine IV continuously on days 4-7, and idarubicin IV over 15 minutes on days 4-6. Patients with residual blasts may receive re-induction treatment beginning on day 28. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
  CONSOLIDATION: Patients receive vorinostat PO TID on days 1-3, cytarabine IV continuously on days 4-6, and idarubicin IV over 15 minutes on days 4-5.
  TRANSPLANT: Patients may undergo an allogeneic transplant after induction therapy or consolidation therapy. (Permanently closed to accrual, effective 6/2/2015) Patients previously randomized to Arm III may continue treatment with or without vorinostat.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic transplant
  Cytarabine: Given IV
  Idarubicin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Vorinostat: Given PO
Period: Overall Study
Arm/Group | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) | Arm II (High-dose Cytarabine, Idarubicin) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin)
Started | 263 | 267 | 224
High Risk Patients | 60 | 61 | 38
High Risk Patients Achieved CR/CRi | 38 | 40 | 29
Known NPM1 Status at Baseline | 169 | 156 | 142
Known Cytogenetic Risk at Baseline | 252 | 250 | 210
Completed | 214 | 206 | 161
Not Completed | 49 | 61 | 63
Not completed — Ineligible | 2 | 6 | 8
Not completed — Adverse Event | 1 | 8 | 8
Not completed — Withdrawal by Subject | 6 | 6 | 5
Not completed — Progression/relapse | 1 | 3 | 0
Not completed — Death | 7 | 14 | 13
Not completed — Other - not protocol specified | 32 | 22 | 24
Not completed — Did not start treatment | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Arm III (Vorinostat, High-dose Cytarabine, Idarubicin): INDUCTION/RE-INDUCTIONI: Patients receive vorinostat PO TID on days 1-3, high-dose cytarabine IV continuously on days 4-7, and idarubicin IV over 15 minutes on days 4-6. Patients with residual blasts may receive re-induction treatment beginning on day 28. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
  CONSOLIDATION: Patients receive vorinostat PO TID on days 1-3, cytarabine IV continuously on days 4-6, and idarubicin IV over 15 minutes on days 4-5.
  TRANSPLANT: Patients may undergo an allogeneic transplant after induction therapy or consolidation therapy. (Permanently closed to accrual, effective 6/2/2015) Patients previously randomized to Arm III may continue treatment with or without vorinostat.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic transplant
  Cytarabine: Given IV
  Idarubicin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Vorinostat: Given PO
- Total: Total of all reporting groups
Arm/Group | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) | Arm II (High-dose Cytarabine, Idarubicin) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin) | Total
Number analyzed (Participants) | 261 | 261 | 216 | 738
Age, Continuous [Median (Full Range); unit: years] | 48.3 [19.2 to 60.8] | 51.5 [18.8 to 60.9] | 48.9 [19.6 to 61.0] | 49.8 [18.8 to 61.0]
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 68 | 65 | 55 | 188
  >= 40 years | 193 | 196 | 161 | 550
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 127 | 102 | 360
  Male | 130 | 134 | 114 | 378
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 22 | 21 | 62
  Not Hispanic or Latino | 226 | 217 | 185 | 628
  Unknown or Not Reported | 16 | 22 | 10 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3 | 6
  Asian | 6 | 4 | 7 | 17
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 19 | 19 | 17 | 55
  White | 218 | 217 | 178 | 613
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 12 | 19 | 11 | 42
Onset of Leukemia [Count of Participants; unit: Participants]
  De novo | 236 | 236 | 193 | 665
  Tx. related/arose from antecededent hem. disease | 25 | 25 | 23 | 73

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: EFS is calculated for all patients from the date of initial registration on study until the first of the following: death from any cause, relapse from remission (CR or CRi) or completion of protocol Induction/Re-Induction therapy without documentation of CR or CRi.
  2-year EFS by arm will be estimated using the Kaplan-Meier method. EFS will be compared between Arm I and Arm III and between Arm II and Arm III using Cox proportional hazards regression.
Time Frame: EFS assessed for up to 5 years, 2 year EFS reported
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) | Arm II (High-dose Cytarabine, Idarubicin) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin)
Number analyzed (Participants) | 261 | 261 | 216
Proportion of participants | 0.36 [0.30 to 0.42] | 0.41 [0.35 to 0.46] | 0.37 [0.30 to 0.43]
Statistical Analysis 1: Comparison: Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) vs Arm III (Vorinostat, High-dose Cytarabine, Idarubicin); Arm I was compared with Arm III using a two-sided test of the null hypothesis (HR=1) at the 0.045 level; Test type: Other; p = 0.84, Regression, Cox; Adjusted for: Age (< 40 vs. >= 40) and Onset of AML (de novo vs. treatment related and/or AML arising from antecedent hematologic disease)
Statistical Analysis 2: Comparison: Arm II (High-dose Cytarabine, Idarubicin) vs Arm III (Vorinostat, High-dose Cytarabine, Idarubicin); Arm II was compared with Arm III using a two-sided test of the null hypothesis (HR=1) at the 0.045 level; Test type: Other; p = 0.42, Regression, Cox; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Rate of Allogeneic HCT
Description: The goal of the transplant objective is to determine whether it is possible to conduct allogeneic HCT on 60% or more of adults with high-risk AML in first complete remission (alternative). If 40% or fewer of high-risk patients in CR can be transplanted, the proposed transplant support system will not be considered feasible. A one-sided binomial test compared to the null transplant rate will be conducted.
Time Frame: Up to 5 years
Population: Eligible patients with high-risk AML who achieved CR or CRi, regardless of treatment arm.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- High Risk Patients in First Complete Remission: This group includes patients from any of the three treatment arms who have high-risk AML (by cytogenetics) and who achieved a complete remission (CR) or complete remission with incomplete blood count recovery (CRi).
Arm/Group | High Risk Patients in First Complete Remission
Number analyzed (Participants) | 107
percentage of patients | 65 [56 to 74]
Statistical Analysis 1: Comparison: High Risk Patients in First Complete Remission; Test type: Other; p < 0.0001, Exact binomial test, 1-sided

3. Secondary Outcome: Disease-free Survival (DFS) Among High Risk Patients
Description: DFS is calculated for patients who have achieved a CR or CRi (complete response with incomplete blood count recovery). DFS will be measured from the date of CR or CRi until relapse from CR or CRi for death from any cause. Observation is censored at the date of last follow-up for patients last known to be alive without report of relapse.
  2-year DFS for high risk patients will be estimated using the Kaplan-Meier method.
Time Frame: DFS assessed for up to 5 years, 2 year DFS reported
Population: Eligible, high risk patients, regardless of treatment arm.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- High Risk Patients: This group includes patients from any of the three treatment arms who have high-risk AML (by cytogenetics).
Arm/Group | High Risk Patients
Number analyzed (Participants) | 159
Proportion of participants | 0.30 [0.21 to 0.39]

4. Secondary Outcome: EFS of Arm I Compared to Arm II
Description: EFS is calculated for all patients from the date of initial registration on study until the first of the following: death from any cause, relapse from remission (CR or CRi) or completion of protocol Induction/Re-Induction therapy without documentation of CR or CRi.
  A two-sided test of the hazard ratio (HR) of 7:3: IA (versus the null hypothesis of HR =1) will be done using a proportional hazards regression model with the stratification factors included as covariates.
  2-year EFS by arm will be estimated using the Kaplan-Meier method.
Time Frame: EFS assessed for up to 5 years, 2 year EFS reported
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) | Arm II (High-dose Cytarabine, Idarubicin)
Number analyzed (Participants) | 261 | 261
Proportion of participants | 0.36 [0.30 to 0.42] | 0.41 [0.35 to 0.46]
Statistical Analysis 1: Comparison: Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) vs Arm II (High-dose Cytarabine, Idarubicin); Arm I was compared with Arm II using a two-sided test of the null hypothesis (HR=1); Test type: Other; p = 0.52, Regression, Cox; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Frequency and Severity of Toxicities
Description: Number of patients with Grade 3-5 adverse events that were possibly, probably or definitely related to study drug are reported by given type of adverse event.
Time Frame: Up to 5 years
Population: Eligible patients who started treatment
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride): INDUCTION/RE-INDUCTION: Patients receive standard dose cytarabine IV continuously on days 1-7 and daunorubicin hydrochloride IV on days 1-3. Patients with residual blasts may receive re-induction treatment beginning on day 15. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
- Arm II (High-dose Cytarabine, Idarubicin): INDUCTION/RE-INDUCTION: Patients receive high dose cytarabine IV continuously on days 1-4 and idarubicin IV over 15 minutes on days 1-3. Patients with residual blasts may receive re-induction treatment beginning on day 28. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
- Arm III (Vorinostat, High-dose Cytarabine, Idarubicin): INDUCTION/RE-INDUCTION: Patients receive vorinostat PO TID on days 1-3, high-dose cytarabine IV continuously on days 4-7, and idarubicin IV over 15 minutes on days 4-6. Patients with residual blasts may receive re-induction treatment beginning on day 28. Patients achieving CR or CRi may proceed to allogeneic HSCT or to consolidation therapy.
Arm/Group | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) | Arm II (High-dose Cytarabine, Idarubicin) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin)
Number analyzed (Participants) | 261 | 259 | 211
Participants
  Abdominal distension | 1 | 0 | 1
  Abdominal infection | 1 | 1 | 1
  Abdominal pain | 4 | 6 | 9
  Acidosis | 1 | 1 | 2
  Acute kidney injury | 2 | 5 | 4
  Adult respiratory distress syndrome | 1 | 3 | 4
  Alanine aminotransferase increased | 12 | 17 | 20
  Alkaline phosphatase increased | 2 | 2 | 1
  Alkalosis | 1 | 1 | 2
  Allergic reaction | 0 | 0 | 2
  Anal hemorrhage | 0 | 0 | 1
  Anal pain | 0 | 1 | 0
  Anal ulcer | 0 | 0 | 1
  Anemia | 158 | 164 | 106
  Anorectal infection | 0 | 0 | 4
  Anorexia | 5 | 16 | 12
  Aspartate aminotransferase increased | 8 | 15 | 12
  Atelectasis | 0 | 0 | 1
  Atrial fibrillation | 0 | 3 | 1
  Atrial flutter | 0 | 1 | 1
  Atrioventricular block complete | 0 | 1 | 0
  Blood and lymphatic system disorders - Other | 1 | 1 | 0
  Blood bilirubin increased | 9 | 15 | 22
  Bone infection | 1 | 0 | 0
  Bone pain | 0 | 1 | 0
  Bronchopulmonary hemorrhage | 1 | 1 | 3
  Bullous dermatitis | 0 | 2 | 0
  CD4 lymphocytes decreased | 1 | 1 | 0
  Cardiac arrest | 1 | 3 | 2
  Cardiac disorders - Other, specify | 1 | 1 | 1
  Cardiac troponin I increased | 0 | 1 | 0
  Catheter related infection | 3 | 7 | 4
  Chills | 1 | 0 | 0
  Chronic kidney disease | 0 | 2 | 0
  Cognitive disturbance | 0 | 0 | 1
  Colitis | 3 | 9 | 5
  Colonic hemorrhage | 2 | 0 | 1
  Colonic perforation | 0 | 0 | 1
  Conduction disorder | 1 | 0 | 0
  Confusion | 0 | 2 | 0
  Conjunctivitis | 1 | 0 | 0
  Constipation | 0 | 1 | 0
  Constrictive pericarditis | 1 | 0 | 0
  Creatinine increased | 1 | 6 | 4
  Death NOS | 1 | 1 | 0
  Dehydration | 1 | 0 | 3
  Dental caries | 1 | 0 | 0
  Device related infection | 1 | 3 | 0
  Diarrhea | 15 | 20 | 38
  Disseminated intravascular coagulation | 2 | 1 | 1
  Dry mouth | 0 | 1 | 0
  Dry skin | 0 | 2 | 0
  Duodenal hemorrhage | 1 | 0 | 0
  Dyspepsia | 1 | 0 | 0
  Dysphagia | 1 | 1 | 0
  Dyspnea | 3 | 7 | 8
  Edema cerebral | 0 | 0 | 1
  Edema limbs | 0 | 3 | 2
  Ejection fraction decreased | 2 | 6 | 4
  Electrocardiogram QT corrected interval prolonged | 0 | 2 | 2
  Encephalopathy | 0 | 1 | 0
  Enterocolitis | 1 | 6 | 5
  Enterocolitis infectious | 1 | 4 | 4
  Epistaxis | 2 | 1 | 2
  Erythema multiforme | 1 | 0 | 0
  Erythroderma | 0 | 0 | 1
  Esophageal hemorrhage | 0 | 0 | 1
  Esophageal pain | 1 | 1 | 0
  Esophagitis | 3 | 2 | 1
  Eye infection | 0 | 1 | 0
  Fatigue | 14 | 18 | 13
  Febrile neutropenia | 152 | 160 | 114
  Fever | 4 | 7 | 6
  GGT increased | 3 | 2 | 4
  Gait disturbance | 0 | 0 | 1
  Gastric hemorrhage | 0 | 2 | 3
  Gastritis | 1 | 0 | 0
  Gastroesophageal reflux disease | 1 | 0 | 0
  Gastrointestinal disorders - Other, specify | 1 | 5 | 1
  General disorders and admin site conditions-Other | 0 | 4 | 1
  Generalized muscle weakness | 2 | 1 | 2
  Genital edema | 0 | 0 | 1
  Glucose intolerance | 1 | 0 | 0
  Gum infection | 1 | 0 | 0
  Headache | 2 | 2 | 4
  Heart failure | 3 | 2 | 3
  Hematoma | 0 | 1 | 0
  Hematuria | 0 | 2 | 0
  Hepatic failure | 1 | 0 | 0
  Hepatic infection | 1 | 1 | 0
  Hepatobiliary disorders - Other, specify | 1 | 0 | 1
  Hyperglycemia | 5 | 12 | 16
  Hyperhidrosis | 1 | 1 | 0
  Hyperkalemia | 0 | 1 | 1
  Hypermagnesemia | 0 | 1 | 0
  Hypernatremia | 0 | 0 | 2
  Hypertension | 7 | 6 | 6
  Hyperuricemia | 0 | 1 | 1
  Hypoalbuminemia | 5 | 8 | 8
  Hypocalcemia | 8 | 17 | 25
  Hypoglycemia | 0 | 0 | 1
  Hypokalemia | 18 | 20 | 24
  Hypomagnesemia | 0 | 1 | 2
  Hyponatremia | 20 | 20 | 9
  Hypophosphatemia | 21 | 31 | 31
  Hypotension | 3 | 12 | 9
  Hypoxia | 2 | 4 | 9
  Ileus | 0 | 1 | 2
  Infections and infestations - Other, specify | 18 | 21 | 14
  Infective myositis | 1 | 0 | 0
  Injury, poison and procedural complications-Other | 1 | 0 | 0
  Intracranial hemorrhage | 0 | 0 | 1
  Investigations - Other, specify | 1 | 6 | 3
  Irregular menstruation | 1 | 0 | 0
  Jejunal obstruction | 0 | 0 | 1
  Kidney infection | 0 | 1 | 0
  Laryngeal edema | 1 | 0 | 0
  Laryngeal mucositis | 0 | 0 | 1
  Left ventricular systolic dysfunction | 2 | 3 | 0
  Leukocytosis | 1 | 1 | 1
  Lipase increased | 0 | 0 | 2
  Lower gastrointestinal hemorrhage | 0 | 1 | 3
  Lung infection | 21 | 22 | 14
  Lymphocyte count decreased | 89 | 107 | 77
  Menorrhagia | 1 | 0 | 0
  Metabolism and nutrition disorders-Other, specify | 1 | 1 | 0
  Middle ear inflammation | 1 | 0 | 0
  Mucosal infection | 1 | 0 | 1
  Mucositis oral | 19 | 18 | 11
  Multi-organ failure | 1 | 3 | 5
  Musculoskeletal and connective tiss disorder-Other | 0 | 1 | 1
  Myalgia | 0 | 0 | 1
  Nausea | 7 | 15 | 5
  Neck edema | 0 | 0 | 1
  Nervous system disorders - Other, specify | 0 | 1 | 0
  Neutrophil count decreased | 141 | 128 | 104
  Non-cardiac chest pain | 1 | 0 | 1
  Oral pain | 5 | 5 | 0
  Pain | 1 | 0 | 0
  Pain in extremity | 1 | 0 | 1
  Palmar-plantar erythrodysesthesia syndrome | 0 | 2 | 1
  Papulopustular rash | 0 | 1 | 0
  Paresthesia | 0 | 0 | 1
  Pericardial effusion | 0 | 0 | 1
  Pericardial tamponade | 0 | 0 | 1
  Periorbital edema | 0 | 1 | 0
  Peripheral sensory neuropathy | 0 | 0 | 1
  Pharyngeal mucositis | 1 | 0 | 0
  Pharyngitis | 1 | 0 | 0
  Platelet count decreased | 175 | 168 | 128
  Pleural effusion | 1 | 0 | 1
  Pneumonitis | 1 | 4 | 2
  Pruritus | 0 | 1 | 1
  Pulmonary edema | 1 | 2 | 5
  Purpura | 0 | 1 | 0
  Rash acneiform | 1 | 1 | 0
  Rash maculo-papular | 11 | 26 | 10
  Rectal hemorrhage | 1 | 0 | 0
  Rectal pain | 1 | 0 | 1
  Renal and urinary disorders - Other, specify | 0 | 1 | 0
  Resp, thoracic and mediastinal disorders - Other | 1 | 3 | 2
  Respiratory failure | 3 | 8 | 14
  Restrictive cardiomyopathy | 1 | 0 | 0
  Salivary duct inflammation | 1 | 0 | 0
  Scrotal infection | 0 | 0 | 1
  Scrotal pain | 0 | 0 | 1
  Seizure | 1 | 0 | 1
  Sepsis | 16 | 26 | 34
  Sinus bradycardia | 0 | 0 | 1
  Sinus tachycardia | 0 | 2 | 2
  Sinusitis | 2 | 0 | 0
  Skin and subcutaneous tissue disorders - Other | 0 | 2 | 1
  Skin infection | 5 | 1 | 4
  Skin ulceration | 0 | 0 | 1
  Small intestinal obstruction | 1 | 0 | 0
  Soft tissue infection | 1 | 0 | 0
  Sore throat | 1 | 2 | 2
  Stomach pain | 1 | 0 | 0
  Stroke | 0 | 1 | 1
  Supraventricular tachycardia | 0 | 1 | 1
  Syncope | 2 | 2 | 3
  Testicular disorder | 0 | 1 | 0
  Thromboembolic event | 1 | 0 | 0
  Thrombotic thrombocytopenic purpura | 3 | 0 | 1
  Tooth infection | 1 | 0 | 0
  Tumor lysis syndrome | 4 | 8 | 9
  Typhlitis | 8 | 14 | 23
  Upper gastrointestinal hemorrhage | 1 | 0 | 1
  Upper respiratory infection | 2 | 1 | 2
  Urinary incontinence | 0 | 0 | 1
  Urinary tract infection | 5 | 2 | 6
  Urine output decreased | 0 | 0 | 1
  Vaginal hemorrhage | 0 | 0 | 2
  Vascular access complication | 0 | 2 | 1
  Vasovagal reaction | 0 | 1 | 1
  Ventricular tachycardia | 0 | 1 | 0
  Vomiting | 3 | 6 | 4
  Weight loss | 2 | 0 | 2
  White blood cell decreased | 156 | 150 | 112
  Wound infection | 1 | 0 | 0

6. Other Pre Specified Outcome: Prevalence of the Mutation NPM1 in Patients on This Study.
Description: To estimate the prevalence of the mutation NPM1 in this patient population.
Time Frame: Baseline
Population: Eligible patients with known NPM1 status at baseline
Measure: Number; unit: percentage of patients
Groups:
- All Arms Combined: This group includes all patients enrolled to the trial, regardless of treatment assignment.
Arm/Group | All Arms Combined
Number analyzed (Participants) | 467
percentage of patients | 33

7. Other Pre Specified Outcome: Prevalence of the Mutations IDH1, IDH2, TET2, DMT3A in Patients on This Study
Description: To estimate the prevalence of these mutations in this patient population.
  This objective will be analyzed as funding allows.
Time Frame: Baseline
Population: There was not sufficient funding to test patients for IDH1, IDH2, TET2, or DMT3A. Therefore, this objective was not completed.
Arm/Group | All Arms Combined
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Cytogenetic Risk Distribution of Patients on This Study
Description: To estimate the cytogenetic risk distribution of patients on this study.
Time Frame: Baseline
Population: Eligible patients with known cytogenetic risk at baseline
Measure: Number; unit: percentage of participants
Arm/Group | All Arms Combined
Number analyzed (Participants) | 712
percentage of participants
  High risk | 22.3
  Intermediate risk | 64.2
  Low risk | 13.5

9. Other Pre Specified Outcome: Overall Survival (OS)
Description: To compare OS between patients who receive standard 7+3 therapy or IA to patients who receive IA + vorinostat.
  OS is calculated for all patients from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
  2-year OS by arm will be estimated using the Kaplan-Meier method.
Time Frame: OS assessed for up to 5 years, 2 year OS reported
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) | Arm II (High-dose Cytarabine, Idarubicin) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin)
Number analyzed (Participants) | 261 | 261 | 216
Proportion of participants | 0.56 [0.50 to 0.62] | 0.59 [0.53 to 0.65] | 0.58 [0.50 to 0.64]

10. Other Pre Specified Outcome: Complete Response (CR) Rate
Description: To compare the complete response rate between patients who receive standard 7+3 therapy or IA to patients who receive IA + vorinostat.
  Complete response is defined as: ANC >= 1,000/mcl, platelet count >= 100,000/mcl, < 5% bone marrow blasts, no Auer rods, no evidence of extramedullary disease (no requirements for marrow cellularity or hemoglobin concentration)
Time Frame: Up to 5 years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) | Arm II (High-dose Cytarabine, Idarubicin) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin)
Number analyzed (Participants) | 261 | 261 | 216
Percentage of participants | 75 [70 to 81] | 80 [74 to 84] | 77 [71 to 83]

11. Other Pre Specified Outcome: Disease-free Survival (DFS)
Description: To compare the disease-free survival (DFS) between patients who receive standard 7+3 therapy or IA to patients who receive IA + vorinostat.
  DFS is calculated for patients who have achieved a CR or CRi (complete response with incomplete blood count recovery) . DFS will be measured from the date of CR or CRi until relapse from CR or CRi for death from any cause. Observation is censored at the date of last follow-up for patients last known to be alive without report of relapse.
  2-year DFS by arm will be estimated using the Kaplan-Meier method.
Time Frame: DFS assessed for up to 5 years, 2 year DFS reported
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) | Arm II (High-dose Cytarabine, Idarubicin) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin)
Number analyzed (Participants) | 261 | 261 | 216
Proportion of participants | 0.48 [0.41 to 0.55] | 0.51 [0.44 to 0.57] | 0.46 [0.38 to 0.54]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Number of patients with adverse events are reported by type of adverse event. All adverse events, regardless of attribution or grade, are reported. Adverse events are reported for eligible patients who started treatment.
Arm/Group | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) | Arm II (High-dose Cytarabine, Idarubicin) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin)
All-Cause Mortality (participants affected / at risk) | 126/261 | 114/259 | 103/211
Serious Adverse Events (participants affected / at risk) | 11/261 | 27/259 | 75/211
Other Adverse Events (participants affected / at risk) | 249/261 | 254/259 | 206/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) (N=261) | Arm II (High-dose Cytarabine, Idarubicin) (N=259) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin) (N=211)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 13
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 4 | 2
Heart failure (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 3
Pericardial tamponade (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 5
Colitis (Gastrointestinal disorders) | 0 | 0 | 6
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 6
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 2
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 2
Jejunal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Typhlitis (Gastrointestinal disorders) | 1 | 0 | 7
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Death NOS (General disorders) | 2 | 1 | 1
Edema limbs (General disorders) | 0 | 0 | 2
Edema trunk (General disorders) | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1
General disorders and admin site conditions - Other (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 2 | 4
Neck edema (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatobiliary disorders-Other (Hepatobiliary disorders) | 1 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Infections and infestations-Other (Infections and infestations) | 0 | 0 | 5
Lip infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 4
Sepsis (Infections and infestations) | 1 | 11 | 17
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 6
Alkaline phosphatase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 5
Blood bilirubin increased (Investigations) | 0 | 1 | 7
Cardiac troponin I increased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 3
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1
Fibrinogen decreased (Investigations) | 0 | 0 | 1
GGT increased (Investigations) | 0 | 0 | 2
INR increased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2
Weight gain (Investigations) | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 6
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1
Edema cerebral (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 2
Ischemia cerebrovascular (Nervous system disorders) | 0 | 0 | 1
Nervous system disorders-Other (Nervous system disorders) | 1 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 3
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 4 | 9
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Genital edema (Reproductive system and breast disorders) | 0 | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 15
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 2 | 8
Thromboembolic event (Vascular disorders) | 0 | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Standard Dose Cytarabine, Daunorubicin Hydrochloride) (N=261) | Arm II (High-dose Cytarabine, Idarubicin) (N=259) | Arm III (Vorinostat, High-dose Cytarabine, Idarubicin) (N=211)
Anemia (Blood and lymphatic system disorders) | 185 | 185 | 137
Febrile neutropenia (Blood and lymphatic system disorders) | 158 | 170 | 120
Sinus bradycardia (Cardiac disorders) | 11 | 9 | 12
Sinus tachycardia (Cardiac disorders) | 44 | 47 | 30
Ear pain (Ear and labyrinth disorders) | 16 | 7 | 2
Blurred vision (Eye disorders) | 15 | 13 | 16
Eye disorders-Other (Eye disorders) | 16 | 15 | 8
Abdominal distension (Gastrointestinal disorders) | 13 | 7 | 11
Abdominal pain (Gastrointestinal disorders) | 59 | 93 | 76
Bloating (Gastrointestinal disorders) | 12 | 16 | 9
Colitis (Gastrointestinal disorders) | 5 | 15 | 10
Constipation (Gastrointestinal disorders) | 80 | 47 | 42
Diarrhea (Gastrointestinal disorders) | 129 | 213 | 157
Dry mouth (Gastrointestinal disorders) | 28 | 19 | 20
Dyspepsia (Gastrointestinal disorders) | 19 | 14 | 22
Dysphagia (Gastrointestinal disorders) | 21 | 17 | 14
Gastroesophageal reflux disease (Gastrointestinal disorders) | 16 | 17 | 14
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 15 | 19 | 11
Hemorrhoids (Gastrointestinal disorders) | 16 | 7 | 17
Mucositis oral (Gastrointestinal disorders) | 95 | 92 | 66
Nausea (Gastrointestinal disorders) | 146 | 181 | 147
Oral hemorrhage (Gastrointestinal disorders) | 14 | 2 | 6
Oral pain (Gastrointestinal disorders) | 30 | 22 | 13
Typhlitis (Gastrointestinal disorders) | 10 | 14 | 18
Vomiting (Gastrointestinal disorders) | 69 | 124 | 93
Chills (General disorders) | 47 | 46 | 37
Edema face (General disorders) | 12 | 13 | 9
Edema limbs (General disorders) | 71 | 89 | 45
Fatigue (General disorders) | 138 | 143 | 105
Fever (General disorders) | 77 | 83 | 55
General disorders and admin site conditions - Other (General disorders) | 16 | 29 | 9
Infusion related reaction (General disorders) | 15 | 13 | 6
Malaise (General disorders) | 7 | 13 | 4
Non-cardiac chest pain (General disorders) | 26 | 20 | 16
Pain (General disorders) | 27 | 34 | 17
Catheter related infection (Infections and infestations) | 6 | 8 | 12
Infections and infestations-Other (Infections and infestations) | 37 | 46 | 31
Lung infection (Infections and infestations) | 32 | 34 | 24
Sepsis (Infections and infestations) | 22 | 20 | 21
Bruising (Injury, poisoning and procedural complications) | 11 | 15 | 9
Activated partial thromboplastin time prolonged (Investigations) | 11 | 19 | 11
Alanine aminotransferase increased (Investigations) | 99 | 109 | 87
Alkaline phosphatase increased (Investigations) | 69 | 70 | 66
Aspartate aminotransferase increased (Investigations) | 89 | 108 | 94
Blood bilirubin increased (Investigations) | 68 | 90 | 72
Creatinine increased (Investigations) | 20 | 32 | 35
INR increased (Investigations) | 36 | 53 | 29
Investigations-Other (Investigations) | 13 | 20 | 11
Lymphocyte count decreased (Investigations) | 98 | 113 | 84
Neutrophil count decreased (Investigations) | 155 | 139 | 112
Platelet count decreased (Investigations) | 185 | 180 | 142
Weight loss (Investigations) | 40 | 37 | 40
White blood cell decreased (Investigations) | 163 | 154 | 121
Anorexia (Metabolism and nutrition disorders) | 81 | 103 | 84
Hyperglycemia (Metabolism and nutrition disorders) | 92 | 98 | 89
Hyperkalemia (Metabolism and nutrition disorders) | 15 | 21 | 11
Hypermagnesemia (Metabolism and nutrition disorders) | 13 | 17 | 14
Hypernatremia (Metabolism and nutrition disorders) | 13 | 16 | 19
Hypoalbuminemia (Metabolism and nutrition disorders) | 127 | 130 | 99
Hypocalcemia (Metabolism and nutrition disorders) | 99 | 109 | 100
Hypoglycemia (Metabolism and nutrition disorders) | 6 | 4 | 11
Hypokalemia (Metabolism and nutrition disorders) | 109 | 127 | 98
Hypomagnesemia (Metabolism and nutrition disorders) | 41 | 49 | 39
Hyponatremia (Metabolism and nutrition disorders) | 93 | 106 | 68
Hypophosphatemia (Metabolism and nutrition disorders) | 71 | 91 | 69
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 29 | 24
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 20 | 15 | 18
Neck pain (Musculoskeletal and connective tissue disorders) | 14 | 6 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 25 | 22
Dizziness (Nervous system disorders) | 34 | 22 | 33
Dysgeusia (Nervous system disorders) | 26 | 38 | 31
Headache (Nervous system disorders) | 74 | 70 | 51
Anxiety (Psychiatric disorders) | 41 | 62 | 35
Confusion (Psychiatric disorders) | 11 | 16 | 10
Depression (Psychiatric disorders) | 19 | 28 | 14
Insomnia (Psychiatric disorders) | 49 | 51 | 39
Acute kidney injury (Renal and urinary disorders) | 9 | 19 | 26
Hematuria (Renal and urinary disorders) | 14 | 17 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 48 | 40
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 55 | 54 | 40
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 35 | 37 | 27
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 14 | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20 | 14 | 12
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 | 17 | 19
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 9
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 11 | 15 | 8
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 7 | 20 | 10
Sore throat (Respiratory, thoracic and mediastinal disorders) | 34 | 18 | 18
Alopecia (Skin and subcutaneous tissue disorders) | 46 | 41 | 46
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 29 | 22
Erythema multiforme (Skin and subcutaneous tissue disorders) | 8 | 13 | 4
Periorbital edema (Skin and subcutaneous tissue disorders) | 6 | 14 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 38 | 58 | 42
Purpura (Skin and subcutaneous tissue disorders) | 11 | 15 | 6
Rash acneiform (Skin and subcutaneous tissue disorders) | 11 | 13 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 94 | 117 | 82
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 29 | 39 | 25
Hypertension (Vascular disorders) | 38 | 54 | 27
Hypotension (Vascular disorders) | 39 | 45 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT01802333/Prot_SAP_000.pdf